CLINICAL TRIAL: NCT02758496
Title: A Chart Review to Evaluate the Safety and Efficacy of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) on Subjects With Autism Spectrum Disorder (ASD)
Brief Title: A Chart Review to Evaluate the Safety and Efficacy of MeRT on Subjects With ASD
Status: Completed | Type: Observational
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: MeRT-016
Record Dates: First submitted 2016-04-15; First posted 2016-05-02 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Autistic Disorder
Keywords: Autism, chart review, transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ASD Subjects: Approximately two hundred (200) male and female subjects of any ethnic background between the ages of 2-20 years old seen at the Brain Treatment Center (BTC) between 2010 and 2015.
  Interventions: Other: MeRT Efficacy Chart Review
- Healthy Controls: Twenty (20) male and female subjects of any ethnic background between the ages of 2-20 years old with 'neurotypical' EEGs will be selected for comparison to the ASD group
  Interventions: Other: MeRT Efficacy Chart Review

INTERVENTIONS:
Other: MeRT Efficacy Chart Review — There will be not intervention. This is a chart review.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) on subjects with Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
This is a retrospective chart review of 200 consecutive charts of subjects ages 2-20 years old seen at the Brain Treatment Center between 2010 and 2015. The review is designed to evaluate the safety and efficacy of Magnetic Electroencephalogram/Electrocardiogram(EEG/ECG)-Guided Resonance Therapy (MeRT) on subjects with Autism Spectrum Disorder (ASD).

ELIGIBILITY:
Inclusion Criteria:

1. Must have completed a baseline EEG at the Brain Treatment Center (BTC)
2. Age between 2 and 20 years old at initial visit
3. Must have a diagnosis of ASD according to the prevailing standard at that time (i.e., Diagnostic and Statistical Manual-IV (DSM-IV)) (ASD Group only)
4. Must have received Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) for more than (5) sessions (ASD Group only)

   Exclusion Criteria:
5. Clinically significant abnormality or clinically significant unstable medical condition during treatment that in the Investigator's judgment may have may limited interpretation of the results.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Two hundred (200) male and female subjects of any ethnic background between the ages of 2-20 years old seen at the Brain Treatment Center between 2010 and 2015. Twenty (20) male and female subjects of any ethnic background between the ages of 2-20 years old with neurotypical EEGs will be selected for comparison to the ASD group.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | Baseline through study completion, an average of 36 months
  Symptom reduction in ASD will be measured using the reduction in the CARS between two time points: Baseline (BL) CARS and Final CARS Evaluation.

SECONDARY OUTCOMES:
Electrophysiological | Baseline through study completion, an average of 36 months
  Changes in quantitative electroencephalogram (qEEG), will be measured with emphasis on the overall changes between two timepoints: BL EEG and Final EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Young Kim, MD, Principal Investigator — Brain Treatment Center
Locations (1):
- Brain Treatment Center, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krakowiak P, Walker CK, Bremer AA, Baker AS, Ozonoff S, Hansen RL, Hertz-Picciotto I. Maternal metabolic conditions and risk for autism and other neurodevelopmental disorders. Pediatrics. 2012 May;129(5):e1121-8. doi: 10.1542/peds.2011-2583. Epub 2012 Apr 9. PMID 22492772
- [Background] Betancur C, Sakurai T, Buxbaum JD. The emerging role of synaptic cell-adhesion pathways in the pathogenesis of autism spectrum disorders. Trends Neurosci. 2009 Jul;32(7):402-12. doi: 10.1016/j.tins.2009.04.003. Epub 2009 Jun 21. PMID 19541375
- [Background] Crespi B, Stead P, Elliot M. Evolution in health and medicine Sackler colloquium: Comparative genomics of autism and schizophrenia. Proc Natl Acad Sci U S A. 2010 Jan 26;107 Suppl 1(Suppl 1):1736-41. doi: 10.1073/pnas.0906080106. Epub 2009 Dec 1. PMID 19955444
- [Background] Stigler KA, S.T., Posey DJ, McDougle CJ, Autism and immune factors: a comprehensive review. Res Autism Spectr Disord, 3(4): p. 840-860.2009.
- [Background] Sudhof TC. Neuroligins and neurexins link synaptic function to cognitive disease. Nature. 2008 Oct 16;455(7215):903-11. doi: 10.1038/nature07456. PMID 18923512
- [Background] Levy SE, Mandell DS, Schultz RT. Autism. Lancet. 2009 Nov 7;374(9701):1627-38. doi: 10.1016/S0140-6736(09)61376-3. Epub 2009 Oct 12. PMID 19819542
- [Background] Just MA, Cherkassky VL, Keller TA, Kana RK, Minshew NJ. Functional and anatomical cortical underconnectivity in autism: evidence from an FMRI study of an executive function task and corpus callosum morphometry. Cereb Cortex. 2007 Apr;17(4):951-61. doi: 10.1093/cercor/bhl006. Epub 2006 Jun 13. PMID 16772313
- [Background] Buie T, Campbell DB, Fuchs GJ 3rd, Furuta GT, Levy J, Vandewater J, Whitaker AH, Atkins D, Bauman ML, Beaudet AL, Carr EG, Gershon MD, Hyman SL, Jirapinyo P, Jyonouchi H, Kooros K, Kushak R, Levitt P, Levy SE, Lewis JD, Murray KF, Natowicz MR, Sabra A, Wershil BK, Weston SC, Zeltzer L, Winter H. Evaluation, diagnosis, and treatment of gastrointestinal disorders in individuals with ASDs: a consensus report. Pediatrics. 2010 Jan;125 Suppl 1:S1-18. doi: 10.1542/peds.2009-1878C. PMID 20048083
- [Background] Happe F, Ronald A. The 'fractionable autism triad': a review of evidence from behavioural, genetic, cognitive and neural research. Neuropsychol Rev. 2008 Dec;18(4):287-304. doi: 10.1007/s11065-008-9076-8. Epub 2008 Oct 28. PMID 18956240
- [Background] Amaral DG, Schumann CM, Nordahl CW. Neuroanatomy of autism. Trends Neurosci. 2008 Mar;31(3):137-45. doi: 10.1016/j.tins.2007.12.005. Epub 2008 Feb 6. PMID 18258309
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Background] Billstedt E, Gillberg IC, Gillberg C. Autism after adolescence: population-based 13- to 22-year follow-up study of 120 individuals with autism diagnosed in childhood. J Autism Dev Disord. 2005 Jun;35(3):351-60. doi: 10.1007/s10803-005-3302-5. PMID 16119476
- [Background] Langstrom N, Grann M, Ruchkin V, Sjostedt G, Fazel S. Risk factors for violent offending in autism spectrum disorder: a national study of hospitalized individuals. J Interpers Violence. 2009 Aug;24(8):1358-70. doi: 10.1177/0886260508322195. Epub 2008 Aug 13. PMID 18701743
- [Background] Posey DJ, Stigler KA, Erickson CA, McDougle CJ. Antipsychotics in the treatment of autism. J Clin Invest. 2008 Jan;118(1):6-14. doi: 10.1172/JCI32483. PMID 18172517
- [Background] Happe F, Ronald A, Plomin R. Time to give up on a single explanation for autism. Nat Neurosci. 2006 Oct;9(10):1218-20. doi: 10.1038/nn1770. PMID 17001340
- [Background] Larsson HJ, Eaton WW, Madsen KM, Vestergaard M, Olesen AV, Agerbo E, Schendel D, Thorsen P, Mortensen PB. Risk factors for autism: perinatal factors, parental psychiatric history, and socioeconomic status. Am J Epidemiol. 2005 May 15;161(10):916-25; discussion 926-8. doi: 10.1093/aje/kwi123. PMID 15870155
- [Background] Geschwind DH. Autism: many genes, common pathways? Cell. 2008 Oct 31;135(3):391-5. doi: 10.1016/j.cell.2008.10.016. PMID 18984147
- [Background] Hultman CM, Sparen P, Cnattingius S. Perinatal risk factors for infantile autism. Epidemiology. 2002 Jul;13(4):417-23. doi: 10.1097/00001648-200207000-00009. PMID 12094096
- [Background] Cheslack-Postava K, Liu K, Bearman PS. Closely spaced pregnancies are associated with increased odds of autism in California sibling births. Pediatrics. 2011 Feb;127(2):246-53. doi: 10.1542/peds.2010-2371. Epub 2011 Jan 10. PMID 21220394
- [Background] Sebat J, Lakshmi B, Malhotra D, Troge J, Lese-Martin C, Walsh T, Yamrom B, Yoon S, Krasnitz A, Kendall J, Leotta A, Pai D, Zhang R, Lee YH, Hicks J, Spence SJ, Lee AT, Puura K, Lehtimaki T, Ledbetter D, Gregersen PK, Bregman J, Sutcliffe JS, Jobanputra V, Chung W, Warburton D, King MC, Skuse D, Geschwind DH, Gilliam TC, Ye K, Wigler M. Strong association of de novo copy number mutations with autism. Science. 2007 Apr 20;316(5823):445-9. doi: 10.1126/science.1138659. Epub 2007 Mar 15. PMID 17363630
- [Background] Marshall CR, Noor A, Vincent JB, Lionel AC, Feuk L, Skaug J, Shago M, Moessner R, Pinto D, Ren Y, Thiruvahindrapduram B, Fiebig A, Schreiber S, Friedman J, Ketelaars CE, Vos YJ, Ficicioglu C, Kirkpatrick S, Nicolson R, Sloman L, Summers A, Gibbons CA, Teebi A, Chitayat D, Weksberg R, Thompson A, Vardy C, Crosbie V, Luscombe S, Baatjes R, Zwaigenbaum L, Roberts W, Fernandez B, Szatmari P, Scherer SW. Structural variation of chromosomes in autism spectrum disorder. Am J Hum Genet. 2008 Feb;82(2):477-88. doi: 10.1016/j.ajhg.2007.12.009. Epub 2008 Jan 17. PMID 18252227
- [Background] Weiss LA, Shen Y, Korn JM, Arking DE, Miller DT, Fossdal R, Saemundsen E, Stefansson H, Ferreira MA, Green T, Platt OS, Ruderfer DM, Walsh CA, Altshuler D, Chakravarti A, Tanzi RE, Stefansson K, Santangelo SL, Gusella JF, Sklar P, Wu BL, Daly MJ; Autism Consortium. Association between microdeletion and microduplication at 16p11.2 and autism. N Engl J Med. 2008 Feb 14;358(7):667-75. doi: 10.1056/NEJMoa075974. Epub 2008 Jan 9. PMID 18184952
- [Background] Ronald A, Happe F, Bolton P, Butcher LM, Price TS, Wheelwright S, Baron-Cohen S, Plomin R. Genetic heterogeneity between the three components of the autism spectrum: a twin study. J Am Acad Child Adolesc Psychiatry. 2006 Jun;45(6):691-699. doi: 10.1097/01.chi.0000215325.13058.9d. PMID 16721319
- [Background] Rogers SJ. What are infant siblings teaching us about autism in infancy? Autism Res. 2009 Jun;2(3):125-37. doi: 10.1002/aur.81. PMID 19582867
- [Background] Filipek PA, Accardo PJ, Baranek GT, Cook EH Jr, Dawson G, Gordon B, Gravel JS, Johnson CP, Kallen RJ, Levy SE, Minshew NJ, Ozonoff S, Prizant BM, Rapin I, Rogers SJ, Stone WL, Teplin S, Tuchman RF, Volkmar FR. The screening and diagnosis of autistic spectrum disorders. J Autism Dev Disord. 1999 Dec;29(6):439-84. doi: 10.1023/a:1021943802493. PMID 10638459
- [Background] Beaudet AL. Autism: highly heritable but not inherited. Nat Med. 2007 May;13(5):534-6. doi: 10.1038/nm0507-534. No abstract available. PMID 17479094
- [Background] Schmitz C, Rezaie P. The neuropathology of autism: where do we stand? Neuropathol Appl Neurobiol. 2008 Feb;34(1):4-11. doi: 10.1111/j.1365-2990.2007.00872.x. Epub 2007 Oct 26. PMID 17971078
- [Background] Piven J, Palmer P, Jacobi D, Childress D, Arndt S. Broader autism phenotype: evidence from a family history study of multiple-incidence autism families. Am J Psychiatry. 1997 Feb;154(2):185-90. doi: 10.1176/ajp.154.2.185. PMID 9016266
- [Background] Weissman JR, Kelley RI, Bauman ML, Cohen BH, Murray KF, Mitchell RL, Kern RL, Natowicz MR. Mitochondrial disease in autism spectrum disorder patients: a cohort analysis. PLoS One. 2008;3(11):e3815. doi: 10.1371/journal.pone.0003815. Epub 2008 Nov 26. PMID 19043581
- [Background] Frye RE, Melnyk S, Macfabe DF. Unique acyl-carnitine profiles are potential biomarkers for acquired mitochondrial disease in autism spectrum disorder. Transl Psychiatry. 2013 Jan 22;3(1):e220. doi: 10.1038/tp.2012.143. PMID 23340503
- [Background] Fournier KA, Hass CJ, Naik SK, Lodha N, Cauraugh JH. Motor coordination in autism spectrum disorders: a synthesis and meta-analysis. J Autism Dev Disord. 2010 Oct;40(10):1227-40. doi: 10.1007/s10803-010-0981-3. PMID 20195737
- [Background] Sigman M, Dijamco A, Gratier M, Rozga A. Early detection of core deficits in autism. Ment Retard Dev Disabil Res Rev. 2004;10(4):221-33. doi: 10.1002/mrdd.20046. PMID 15666338
- [Background] Sigman M, Spence SJ, Wang AT. Autism from developmental and neuropsychological perspectives. Annu Rev Clin Psychol. 2006;2:327-55. doi: 10.1146/annurev.clinpsy.2.022305.095210. PMID 17716073
- [Background] Iacoboni M, Dapretto M. The mirror neuron system and the consequences of its dysfunction. Nat Rev Neurosci. 2006 Dec;7(12):942-51. doi: 10.1038/nrn2024. Epub 2006 Nov 8. PMID 17115076
- [Background] Association, A.P., Diagnostic and statistical manual of mental disorders; DSM-IV. Vol. 4th. 2000.
- [Background] Johnson CP, Myers SM; American Academy of Pediatrics Council on Children With Disabilities. Identification and evaluation of children with autism spectrum disorders. Pediatrics. 2007 Nov;120(5):1183-215. doi: 10.1542/peds.2007-2361. Epub 2007 Oct 29. PMID 17967920
- [Background] Becker KG. Male gender bias in autism and pediatric autoimmunity. Autism Res. 2012 Apr;5(2):77-83. doi: 10.1002/aur.1227. Epub 2012 Mar 17. PMID 22431266
- [Background] Schopler E, Reichler RJ, DeVellis RF, Daly K. Toward objective classification of childhood autism: Childhood Autism Rating Scale (CARS). J Autism Dev Disord. 1980 Mar;10(1):91-103. doi: 10.1007/BF02408436. No abstract available. PMID 6927682
- [Background] Ozonoff S, Goodlin-Jones BL, Solomon M. Evidence-based assessment of autism spectrum disorders in children and adolescents. J Clin Child Adolesc Psychol. 2005 Sep;34(3):523-40. doi: 10.1207/s15374424jccp3403_8. PMID 16083393
- [Background] Schopler E, v.B.M., Wellman GJ, Love SR, CARS2 Childhood Autism Rating Scale, second edition. WPS Publishing: Torrance, CA. 2010.
- [Background] Helt M, Kelley E, Kinsbourne M, Pandey J, Boorstein H, Herbert M, Fein D. Can children with autism recover? If so, how? Neuropsychol Rev. 2008 Dec;18(4):339-66. doi: 10.1007/s11065-008-9075-9. Epub 2008 Nov 14. PMID 19009353
- [Background] Rogers SJ, Vismara LA. Evidence-based comprehensive treatments for early autism. J Clin Child Adolesc Psychol. 2008 Jan;37(1):8-38. doi: 10.1080/15374410701817808. PMID 18444052
- [Background] Seltzer MM, Shattuck P, Abbeduto L, Greenberg JS. Trajectory of development in adolescents and adults with autism. Ment Retard Dev Disabil Res Rev. 2004;10(4):234-47. doi: 10.1002/mrdd.20038. PMID 15666341
- [Background] Pickett E, Pullara O, O'Grady J, Gordon B. Speech acquisition in older nonverbal individuals with autism: a review of features, methods, and prognosis. Cogn Behav Neurol. 2009 Mar;22(1):1-21. doi: 10.1097/WNN.0b013e318190d185. PMID 19372766
- [Background] Magiati I, Charman T, Howlin P. A two-year prospective follow-up study of community-based early intensive behavioural intervention and specialist nursery provision for children with autism spectrum disorders. J Child Psychol Psychiatry. 2007 Aug;48(8):803-12. doi: 10.1111/j.1469-7610.2007.01756.x. PMID 17683452
- [Background] Fountain C, Winter AS, Bearman PS. Six developmental trajectories characterize children with autism. Pediatrics. 2012 May;129(5):e1112-20. doi: 10.1542/peds.2011-1601. Epub 2012 Apr 2. PMID 22473372
- [Background] MM, S., EEG Waves Classifier using wavelet Transform and Fourier Transform. International Journal of Medical, Pharmaceutical Science and Engineering, 1(3): p. 77 - 82. 2007.
- [Background] Roberts TP, Schmidt GL, Egeth M, Blaskey L, Rey MM, Edgar JC, Levy SE. Electrophysiological signatures: magnetoencephalographic studies of the neural correlates of language impairment in autism spectrum disorders. Int J Psychophysiol. 2008 May;68(2):149-60. doi: 10.1016/j.ijpsycho.2008.01.012. Epub 2008 Feb 12. PMID 18336941
- [Background] Kikuchi M, Yoshimura Y, Shitamichi K, Ueno S, Hirosawa T, Munesue T, Ono Y, Tsubokawa T, Haruta Y, Oi M, Niida Y, Remijn GB, Takahashi T, Suzuki M, Higashida H, Minabe Y. A custom magnetoencephalography device reveals brain connectivity and high reading/decoding ability in children with autism. Sci Rep. 2013;3:1139. doi: 10.1038/srep01139. Epub 2013 Jan 25. PMID 23355952
- [Background] Kondacs A, Szabo M. Long-term intra-individual variability of the background EEG in normals. Clin Neurophysiol. 1999 Oct;110(10):1708-16. doi: 10.1016/s1388-2457(99)00122-4. PMID 10574286
- [Background] Salinsky MC, Oken BS, Morehead L. Test-retest reliability in EEG frequency analysis. Electroencephalogr Clin Neurophysiol. 1991 Nov;79(5):382-92. doi: 10.1016/0013-4694(91)90203-g. PMID 1718711
- [Background] Jin Y, R.A., Thai TM, Huang Y, Therapeutic application of transcranial magnetic stimulation in autism spectrum disorders. Autism Sci Digest, 3: p. 75-79.2010.
- [Background] Jin Y, Potkin SG, Kemp AS, Huerta ST, Alva G, Thai TM, Carreon D, Bunney WE Jr. Therapeutic effects of individualized alpha frequency transcranial magnetic stimulation (alphaTMS) on the negative symptoms of schizophrenia. Schizophr Bull. 2006 Jul;32(3):556-61. doi: 10.1093/schbul/sbj020. Epub 2005 Oct 27. PMID 16254067
- [Background] Klimesch W. An algorithm for the EEG frequency architecture of consciousness and brain body coupling. Front Hum Neurosci. 2013 Nov 12;7:766. doi: 10.3389/fnhum.2013.00766. eCollection 2013. No abstract available. PMID 24273507
- [Background] Melkerson, M., Special Premarket 510(k) Notification for NeuroStar® TMS Therapy System for Major Depressive Disorder. Food and Drug Administration. 2008.
- [Background] V, K., Letter to Brainsway Ltd:510K summary Brainsway Deep TMS system. Office of Device Evaluation, Center for Devices and Radiological Health, Food and Drug Administration. 2013.
- [Background] Release, F.N., FDA allows marketing of first device to relieve migraine headache pain: Cerena Transcranial Magnetic stimulation device. http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm378608.htm. 2013.
- [Background] Jasper H, S.P., Bradley C, Electroencephalographic analyses of behavior problem children. Am J Psychiatry, 95: p. 641. 1938.
- [Background] Matsuura M, Okubo Y, Toru M, Kojima T, He Y, Hou Y, Shen Y, Lee CK. A cross-national EEG study of children with emotional and behavioral problems: a WHO collaborative study in the Western Pacific Region. Biol Psychiatry. 1993 Jul 1-15;34(1-2):59-65. doi: 10.1016/0006-3223(93)90257-e. PMID 8373939
- [Background] Jeong J. EEG dynamics in patients with Alzheimer's disease. Clin Neurophysiol. 2004 Jul;115(7):1490-505. doi: 10.1016/j.clinph.2004.01.001. PMID 15203050
- [Background] Locatelli T, Cursi M, Liberati D, Franceschi M, Comi G. EEG coherence in Alzheimer's disease. Electroencephalogr Clin Neurophysiol. 1998 Mar;106(3):229-37. doi: 10.1016/s0013-4694(97)00129-6. PMID 9743281
- [Background] Loo SK, Makeig S. Clinical utility of EEG in attention-deficit/hyperactivity disorder: a research update. Neurotherapeutics. 2012 Jul;9(3):569-87. doi: 10.1007/s13311-012-0131-z. PMID 22814935
- [Background] Monastra VJ, Lubar JF, Linden M, VanDeusen P, Green G, Wing W, Phillips A, Fenger TN. Assessing attention deficit hyperactivity disorder via quantitative electroencephalography: an initial validation study. Neuropsychology. 1999 Jul;13(3):424-433. doi: 10.1037/0894-4105.13.3.424. PMID 10447303
- [Background] Barry RJ, Johnstone SJ, Clarke AR. A review of electrophysiology in attention-deficit/hyperactivity disorder: II. Event-related potentials. Clin Neurophysiol. 2003 Feb;114(2):184-98. doi: 10.1016/s1388-2457(02)00363-2. PMID 12559225
- [Background] Snyder SM, Hall JR. A meta-analysis of quantitative EEG power associated with attention-deficit hyperactivity disorder. J Clin Neurophysiol. 2006 Oct;23(5):440-55. doi: 10.1097/01.wnp.0000221363.12503.78. PMID 17016156
- [Background] Ogrim G, Kropotov J, Hestad K. The quantitative EEG theta/beta ratio in attention deficit/hyperactivity disorder and normal controls: sensitivity, specificity, and behavioral correlates. Psychiatry Res. 2012 Aug 15;198(3):482-8. doi: 10.1016/j.psychres.2011.12.041. Epub 2012 Mar 16. PMID 22425468
- [Background] Spence SJ, Schneider MT. The role of epilepsy and epileptiform EEGs in autism spectrum disorders. Pediatr Res. 2009 Jun;65(6):599-606. doi: 10.1203/PDR.0b013e31819e7168. PMID 19454962
- [Background] Wang J, Barstein J, Ethridge LE, Mosconi MW, Takarae Y, Sweeney JA. Resting state EEG abnormalities in autism spectrum disorders. J Neurodev Disord. 2013 Sep 16;5(1):24. doi: 10.1186/1866-1955-5-24. PMID 24040879
- [Background] Lansbergen MM, Arns M, van Dongen-Boomsma M, Spronk D, Buitelaar JK. The increase in theta/beta ratio on resting-state EEG in boys with attention-deficit/hyperactivity disorder is mediated by slow alpha peak frequency. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jan 15;35(1):47-52. doi: 10.1016/j.pnpbp.2010.08.004. Epub 2010 Aug 13. PMID 20713113
- [Background] Lansbergen MM, van Dongen-Boomsma M, Buitelaar JK, Slaats-Willemse D. ADHD and EEG-neurofeedback: a double-blind randomized placebo-controlled feasibility study. J Neural Transm (Vienna). 2011 Feb;118(2):275-84. doi: 10.1007/s00702-010-0524-2. Epub 2010 Dec 17. PMID 21165661